CLINICAL TRIAL: NCT03255668
Title: Haematotoxicity in Maintenance Therapy of Children With Acute Lymphoblastic Leukemia: Focus on Genotyping and Phenotyping of Mercaptopurine
Brief Title: Hematotoxicity in Maintenance Therapy of Children With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dewi Selvina Rosdiana, Medical Doctor, MSc, Indonesia University
Other Study IDs: IndonesiaFKUI
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Mercaptopurine Adverse Reaction; Leukemia, Lymphoblastic
Keywords: Mercaptopurine, acute lymphoblastic leukemia, hematotoxicity
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Subjects who are recruited in this study are LLA patient, who are treated for routine control to Cipto Mangunkusumo Hospital, who meet the inclusion criteria and do not meet the exclusion criteria.

DETAILED DESCRIPTION:
On the day of the control patient, (usually the patient is asked for routine control at week 3 on mercaptopurin) routine blood tests are performed. Patients and parents were given an explanation of this study. If patients and parents are willing to take part in the study, they are asked to sign informed consent. Patients who meet the inclusion criteria and do not meet the exclusion criteria, are recorded for demographic data and 5 ml of blood taking. The blood is directly divided into three, 2 mL for hematologic examination and albumin level, 1 mL for genotyping, and 2 mL for examination of drug levels. Routine hematologic examination and albumin levels were performed in the Cipto Mangunkusumo hospital laboratory. For genotypic examination, blood samples were stored at -80C, until they were used for analysis. For examination of the drug levels the blood sample is centrifuged and the erythrocyte preparation is then stored at -80C, until it is used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia (ALL) patients, 1 until 18 years old, male or female, who come to Cipto Mangunkusumo Hospital, Jakarta, Indonesia
* Received 6MP chemotherapy at least 1 month maintenance phase
* Received maintenance phase treatment regimen
* Willing to participate in research, signed informed consent and obtained parental consent to participate in research

Exclusion Criteria:

* Patients are experiencing severe infections
* Patients receiving colony stimulating factor (CSF), allopurinol, mesalazine, olsalazine, and sulfasalazine

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with LLA who received 6-MP chemotherapy in the maintenance phase, who come to RSCM, and who meets the inclusion criteria and does not meet the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Hematotoxicity in Maintenance Therapy of Children With Acute Lymphoblastic Leukemia, the relationship the event with genotyping and phenotyping | August 2017 - May 2018
  Haematology data (hemoglobin, leukocites, platelets, absolute neutrophil count), TPMT genotyping, and blood concentration of 6-meMP and 6-TGN (=phenotyping).

SECONDARY OUTCOMES:
other Factors that can influence the incidence of hematotoxicity | July 2017 - May 2018
  relaps risk stratification (High risk or standard risk), nutrition status,and albumin levels

CONTACTS AND LOCATIONS:
Overall Officials: Rianto Setiabudy, Professor, Study Director — Department of Pharmacology and therapeutic, FMUI; Djajadiman Gatot, Professor, Study Chair — Department of Pediatric
Locations (1):
- Cipto Mangunkusomo hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03255668/Prot_SAP_ICF_000.pdf